CLINICAL TRIAL: NCT04068870
Title: Modification of an Evidence-based Family Planning Intervention for a New Target Population: Postpartum Women in Nakaseke District, Uganda - Pilot Phase, Two Arm
Brief Title: Testing a Modified Family Planning Intervention for Postpartum Women in Uganda
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: African Community Center for Social Sustainability (Unknown)
Responsible Party: Principal Investigator, Sarah Heil, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UGPPFP
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contraceptive management program (Experimental)
  Interventions: Behavioral: Contraceptive management program
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Contraceptive management program — The contraceptive management program will consist of two components: (1) the World Health Organization's contraception protocol and (2) incentivized visits.
  Arms: Contraceptive management program

SUMMARY:
The purpose of this study is to test whether offering incentives to encourage women to attend one-on-one family planning education sessions and offering free, onsite prescription contraceptive methods increases use and continuation of prescription contraception among postpartum women in Uganda. This intervention is modified from one that has been effective outside of Uganda.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* Not planning on getting pregnant in the next 4 months
* Less than 3 months postpartum
* No history of tubal ligation or hysterectomy
* No recent prescription contraceptive use (no pill, intrauterine device or implant use in the past 7 days or injection use in the past 3 months)
* Medically eligible to use prescription contraceptives
* Bringing baby to immunization clinic for the first time

Exclusion Criteria:

* Failure to meet the aforementioned inclusion criteria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Period prevalence use of a prescription contraceptive | 6 months after delivery
  Period prevalence use of a prescription contraceptive

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Heil, PhD, Principal Investigator — University of Vermont
Locations (1):
- Nakaseke District Hospital, Nakaseke, Uganda